CLINICAL TRIAL: NCT02924532
Title: Diagnostic Value of Immediate Postoperative Dose of Parathyroid Hormone as a Marker for the Occurrence of Hypoparathyroidism After Total Thyroidectomy: A Retrospective Observational Study
Brief Title: Postoperative Dose of Parathyroid Hormone as a Marker for the Occurrence of Hypoparathyroidism After Total Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/BL-01
Record Dates: First submitted 2016-09-13; First posted 2016-10-05 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-09

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with total thiroidectomy
  Interventions: Biological: immediate post operative bioassay of Parathyroid Hormone

INTERVENTIONS:
Biological: immediate post operative bioassay of Parathyroid Hormone

SUMMARY:
The main objective of this study is to establish an optimal threshold Early parathormon (PTH) assay in order to exclude hypoparathyroidism , that is to say to obtain a negative predictive value of hypoparathyroidism highest possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively operated on between February 1, 2012 and December 1, 2013
* Total thyroidectomy +/- lymphadenectomy
* Respect of clinicobiological protocol presented above
* The ( the ) patient ( e) was informed ( e) on the implementation of the study 's objectives, constraints and patient rights
* The ( the ) patient ( e) is under ( e) at least 18 years

Exclusion Criteria:

* The ( the ) patient ( e) is under guardianship, curatorship or under guard saves justice
* It is not possible to give to ( the ) patient ( e) informed information
* History of cervical radiotherapy
* Previous history of dysfunction of the parathyroid glands
* Previous history of surgery of the parathyroid glands
* A history of kidney failure or hepatocellular
* History of osteomalacia or Paget's disease
* unhealed cancer antecedent
* History of sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients underwent total thyroidectomy from 1 February 2012 to 1 December 2013 at the Nîmes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-02; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the presence/absence of hypoparathyroidism | day 1
  hypoparathyroidism is defined as: corrected serum calcium Day 1 <1.90 and / or symptoms of hypocalcemia (cramps, tingling of the extremities and peri-oral) to Day 1 authenticated by a VAS score> 3.

REFERENCES:
- [Result] Galy-Bernadoy C, Lallemant B, Chambon G, Pham HT, Reynaud C, Alovisetti C, Bonduelle Q, Guedj AM, Lumbroso S, De Brauwere DP. Parathyroid Hormone Assays following Total Thyroidectomy: Is There a Predictive Value? Eur Thyroid J. 2018 Jan;7(1):34-38. doi: 10.1159/000484689. Epub 2017 Dec 7. PMID 29594052